CLINICAL TRIAL: NCT00702819
Title: Phase 1 Trial of Pan-VEGF Blockade for the Treatment of Retinopathy of Prematurity
Brief Title: Pan-VEGF Blockade for the Treatment of Retinopathy of Prematurity
Acronym: BLOCK-ROP
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low enrollment due to the stringent enrollment criteria. Unable to answer study questions
Sponsor: Vision Research Foundation (Other)
Responsible Party: Michael T. Trese, MD, Vision Research Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IND # 100,633; IND # 100,633
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2008-06

CONDITIONS: Retinopathy of Prematurity
Keywords: Pan-Vascular Endothelial Growth Factor Blockade; Safety
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bevacizumab — Dosage of 0.75mg/0.03ml injectable, one time only.
  Other Names: Avastin

SUMMARY:
Retinopathy of Prematurity (ROP) is a leading cause of blindness in children in developed countries around the world, and an increasing cause of blindness in developing countries.

The retina lines the inside of the eye. It functions as "film" within the camera which is the eye. When an infant is born prematurely, the vascular network necessary to nourish the retina has not fully developed. As a consequence, in some infants abnormal vessels proliferate instead of the normal ones - a condition known as ROP. The abnormal vessels carry scar tissue along with them, and may lead to retinal detachment and blindness if the eye is not treated.

The Multicenter Trial of Cryotherapy for Retinopathy of Prematurity (CRYO-ROP) Study demonstrated that ablation of the peripheral avascular retina reduced the risk of poor structural and visual outcome due to retinal distortion or detachment in ROP (1980's). The ablated retina is not functional and is not amenable to regeneration.

Peripheral retinal ablation is not universally effective in fostering regression of ROP. This is particularly true for an aggressive form of ROP (aggressive posterior ROP, or APROP) which typically afflicts profoundly premature and infirm neonates. In this subset of infants, progression of ROP to bilateral retinal detachment and blindness occurs despite timely and complete peripheral retinal laser ablation.

Rationale The development of ROP is largely dependent on vascular endothelial growth factor (VEGF). When an infant is born prematurely the relatively hyperoxic environment the baby is introduced to shuts down the production of VEGF. Retinal maturation is delayed. Subsequently, at a time when intraocular VEGF levels would normally be declining late in the third trimester of pregnancy, abnormally high levels of VEGF are seen due to large areas of avascular retina and associated tissue hypoxia.

The availability of FDA-approved drugs for anti-VEGF treatment renders it possible to treat such eyes off-label. Available drugs include pegaptanib sodium (Macugen) for partial blockage of VEGF-A, or drugs such as ranibizumab (Lucentis) and bevacizumab (Avastin), which cause complete blockage of VEGF-A.

As VEGF is required in the developing retina for normal angiogenesis, and our goal is not to penetrate tissue, but to block the excessive levels of VEGF trapped within the overlying vitreous which is responsible for the abnormal vasculature in ROP.

For purposes of this study the investigators have chosen bevacizumab (Avastin), which will: a) attain complete blockage (vs. Macugen) of intravitreal VEGF-A, and; b) which is limited in its ability to penetrate tissues because it is a full antibody (vs. Lucentis, an antibody fragment specifically designed for better tissue penetration), and is more likely to restore VEGF homeostasis within the developing retina.

ELIGIBILITY:
Eligibility criteria

* Premature newborn infants with bilateral progressive APROP despite complete peripheral retinal ablation.

Inclusion Criteria:

* Inborn babies at participating NICUs (must meet inclusion criteria 3 through 7)
* Outborn babies transferred to participating NICU (must meet inclusion criteria 3 through 7)
* Aggressive posterior ROP
* Adequate/appropriate laser ablation
* Failed standard laser treatment (persistent Plus or recurrent Plus at a minimum of 1 week post-laser)
* Post-menstrual age less than 36 weeks
* Post-menstrual age greater than 30 weeks

Exclusion Criteria:

* Fatal systemic anomaly
* An ocular anomaly of one or both eyes affecting the retina or choroid
* An ocular anomaly precluding use of the RetCam (eg: microphthalmia)
* Neonatologist feels inclusion will unduly challenge the infant
* Refusal of initial consent
* Refusal of subsequent evaluation
* Media opacity precluding fundus visualization (eg: cataract)
* Any ocular or periocular infection(s)

Ages: 30 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The primary aim is to evaluate the safety of Bevacizumab (Avastin) administered in a single dose into the vitreous cavity. | Weekly

SECONDARY OUTCOMES:
The secondary therapeutic study aim is to determine the efficacy of treatment with Bevacizumab (Avastin) for improving structural outcome without surgical intervention. | Weekly

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Trese, MD, Study Chair — Vision Research Foundation
Locations (11):
- United States (10):
  - Childrens Hospital, Los Angeles, California
  - Jules Stein Eye Center, Los Angeles, California
  - California Vitreoretinal Center, Menlo Park, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - Emory Eye Center, Atlanta, Georgia
  - Children's Hospital / Dept. Ophthalmology, Boston, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - University of North Carolina/Ophthalmology, Chapel Hill, North Carolina
  - University of Pennsylvania/Scheie Eye Institute, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
- Calgary Health, Calgary, Alberta, Canada

REFERENCES:
- [Background] Bakri SJ, Snyder MR, Pulido JS, McCannel CA, Weiss WT, Singh RJ. Six-month stability of bevacizumab (Avastin) binding to vascular endothelial growth factor after withdrawal into a syringe and refrigeration or freezing. Retina. 2006 May-Jun;26(5):519-22. doi: 10.1097/01.iae.0000225354.92444.7a. PMID 16770257